CLINICAL TRIAL: NCT02683850
Title: Influence of an Omega-3 SPM Supplement on Quality of Life
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Metagenics, Inc. (Industry)
Responsible Party: Principal Investigator, Ryan Bradley, Assistant Director of Research, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 091515-B
Record Dates: First submitted 2016-01-31; First posted 2016-02-17 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 SPM (Experimental): Intervention: Study participants will be instructed to take 3 Omega-3 SPM™ softgel supplements in the morning and 3 Omega-3 SPM™ soft gel supplements in the evening for two weeks.
  At weeks two participants whose PROMIS-43 Pain Intensity score indicates a reduction in pain levels weeks, will take 2 Omega-3 SPM™ soft gel supplements in the morning and 2 in the evening for the remaining 2 weeks of the study.
  Participants whose PROMIS-43 Pain Intensity score remained the same after two weeks, or increased will take 4 Omega-3 SPM™ soft gel supplements in the morning and 4 SPM™ softgels in the evening for the remaining two weeks of the study.
  Interventions: Dietary Supplement: Omega-3 SPM™ softgel

INTERVENTIONS:
Dietary Supplement: Omega-3 SPM™ softgel — This four week, prospective, non-randomized, open-label study is assessing the impact on quality of life from taking an Omega-3 SPM™ softgel supplement in adults with pain symptoms at screening of 4 or higher on the PROMIS-43 Profile - Pain Intensity subscale.

SUMMARY:
This prospective, non-randomized, open-label study will assess if taking an Omega-3 SPM™ soft gel supplement for four weeks will increase the quality of life in adults with chronic pain.

DETAILED DESCRIPTION:
One third of the America population is affected by chronic pain. The societal costs associated with chronic pain is up to $635 billion dollars annually. Prescribed pain medications may have negative side effects, or cause addictions. Having alternative treatments that can reduce inflammation and the side effects associated with chronic pain may improve the quality of life for millions.

This prospective, non-randomized, open-label study will assess if taking an Omega-3 SPM™ soft gel supplement for four weeks will increase the quality of life in adults with chronic pain. SPM™ softgels are a dietary supplement intended to reduce pain and inflammation. Up to 40 men and women with chronic pain will be recruited. Outcome measures will be collected at baseline, 2 weeks, and 4 weeks with a primary endpoint of 4 weeks. The primary outcomes of this pilot study include questionnaires to assess quality of life. Exploratory outcomes assess safety and tolerability, changes in anxiety and depression as well as levels of pain, and blood markers associated with inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70
* Body mass index 19 kg/m2 - 40 kg/m2
* Have had chronic pain lasting 3 months or longer
* Have moderate to severe pain as define by an average level of pain score of greater than or equal to a 4 on the PROMIS-43 Profile - Pain Intensity subscale
* Willing to have blood drawn three times
* Maintained stable medications, dietary supplements and therapies for pain for at least 30 days and willing to continue the same therapies and not add new therapies for the duration of the study unless medically advised to do so
* Able to follow study protocol and attend visits at the clinical practices associated with Clinical Investigator
* Able to speak, read and understand English

Exclusion Criteria:

* Initiation of or changes in use of fish oil supplements, krill oil supplements, omega 3 supplements, or omega 3-based drugs (Lovaza®, etc.) within the past 3 months
* Initiation of new pain medications and non-steroidal anti-inflammatory drugs NSAIDS within the past month such as [aspirin, ibuprofen (Advil®, Motrin®, Nuprin®), acetaminophen (Tylenol®), naproxen (Aleve®, Naprosyn®), codeine (Vicodin®), morphine (Dilaudid®), oxycodone (OxyContin®, Percocet®) fentanyl (Duragesic®) and COX-2 inhibitors, Celebrex®)
* Currently taking:

  * Medication to reduce the tendency to form blood clots such as [warfarin, jantoven (Coumadin®); dabigatran (Pradaxa®); rivaroxaban, (Xarelto®); apixaban (Eliquis®)]
  * Statin use for cholesterol reduction such as [atorvastatin (Lipitor®), fluvastatin (Lescol®), lovastatin (Mevacor®, Altocor®), pitavastatin (Livalo®), pravastatin (Pravachol®), rosuvastatin (Crestor®) or simvastatin (Zocor®)] (not including Red Yeast Rice if also supplementing with CoQ10)
  * Corticosteroids such as [prednisone, dexamethasone, prednisolone (Orapred®, Prelone®, Pediapred®), methylprednisolone (Medrol®)] (not including topical corticosteroids for dermatological conditions or nasally inhaled for asthma, rhinitis or sinusitis)
  * Daily aspirin >325 mg per day (not including low dose aspirin therapy of 81 mg - 325 mg per day)
* Other medications and supplements to be evaluated by the investigators on a case-by-case basis
* Steroid injections, Prolotherapy, or other injections into a ligament, tendon, joint or muscle during the past month or initiation or continuation of therapy injections during the course of the study.
* Present or past history of any of the following:

  * Inflammatory disease (e.g. rheumatoid arthritis, autoimmune disease, Crohn's disease, diverticulitis, viral hepatitis, ulcerative colitis, systemic lupus, Parkinson's disease, Alzheimer's, ankylosing spondylitis)
  * Blood clot disorder (e.g., phlebitis)
  * Diabetes (self-report; includes Type I and Type II Diabetes but does not include a history of Gestational Diabetes during pregnancy)
  * Cancer within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
  * Cardiovascular disease within the last year, including but not limited to: myocardial infarction, stroke, congestive heart failure (CHF)
  * Kidney failure or liver failure
* Current active pelvic inflammatory disease, urinary tract infection or a kidney infection
* Women who are lactating, pregnant or planning pregnancy within the next six months
* Difficulty or aversion to swallowing soft gels, capsules, tablets or pills
* Known intolerance or allergy to fish oils
* Upon administering the NCNM Adverse Event Monitoring form at screening, a sign or symptom of Grade 3 (severe or medically significant but not immediately life-threatening) or higher is reported
* Currently participating in another research study or participated in another study within the last month

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life through PROMIS-43 | Four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on quality of life in a chronic pain population using the PROMIS-43 Profile (including PROMIS-43 subscales addressing physical function, fatigue, and sleep disturbance, ability to participate in social roles and activities).
Quality of Life ACPA | Four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on quality of life in a chronic pain population using American Chronic Pain Association's Quality of Life Scale.

OTHER OUTCOMES:
ncidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on safety and tolerability will be monitored by changes in multi-system symptoms using the NCNM Adverse Event Monitoring Form.
Depression and Anxiety PHQ-9 | four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on changes in depression and anxiety determined using the PHQ-9
Depression and Anxiety GAD-7 | four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on changes in depression and anxiety determined using the GAD-7
Depression and Anxiety PROMIS-43 | four weeks
  To assess the effect of 4 weeks of treatment with a SPM supplement on changes in depression and anxiety determined using the PROMIS-43 Profile
Pain | four weeks
  Changes in pain levels, pain symptoms, pain relief, physical function, pain interference, and pain intensity and pain quality determined using the Brief Pain Inventory
Pain | Four weeks
  Changes in physical function, pain interference, and pain intensity the PROMIS-43 Profile subscales
Patient Satisfaction PSS | four weeks
  Patient satisfaction and impression of change determined using the PSS
Patient Satisfaction PGIC | four weeks
  Patient satisfaction and impression of change determined using the PGIC
Pain medication usage | four weeks
  Changes in the use of pain medications determined using the case report form
hs-CRP | four weeks
  Changes in inflammatory biomarkers assessed by high-sensitivity C-reactive protein (hs-CRP)
ESR | four weeks
  Changes in inflammatory biomarkers assessed by erythrocyte sedimentation rate (ESR)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams DI, Dolor R, Roberts R, Pechura C, Dusek J, Amoils S, Amoils S, Barrows K, Edman JS, Frye J, Guarneri E, Kligler B, Monti D, Spar M, Wolever RQ. The BraveNet prospective observational study on integrative medicine treatment approaches for pain. BMC Complement Altern Med. 2013 Jun 24;13:146. doi: 10.1186/1472-6882-13-146. PMID 23800144
- [Background] Ussai S, Miceli L, Pisa FE, Bednarova R, Giordano A, Della Rocca G, Petelin R. Impact of potential inappropriate NSAIDs use in chronic pain. Drug Des Devel Ther. 2015 Apr 9;9:2073-7. doi: 10.2147/DDDT.S80686. eCollection 2015. PMID 25926717
- [Background] Reuben DB, Alvanzo AA, Ashikaga T, Bogat GA, Callahan CM, Ruffing V, Steffens DC. National Institutes of Health Pathways to Prevention Workshop: the role of opioids in the treatment of chronic pain. Ann Intern Med. 2015 Feb 17;162(4):295-300. doi: 10.7326/M14-2775. PMID 25581341
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Maroon JC, Bost JW. Omega-3 fatty acids (fish oil) as an anti-inflammatory: an alternative to nonsteroidal anti-inflammatory drugs for discogenic pain. Surg Neurol. 2006 Apr;65(4):326-31. doi: 10.1016/j.surneu.2005.10.023. PMID 16531187
- [Background] Serhan CN. Pro-resolving lipid mediators are leads for resolution physiology. Nature. 2014 Jun 5;510(7503):92-101. doi: 10.1038/nature13479. PMID 24899309
- [Background] Serhan CN, Chiang N, Van Dyke TE. Resolving inflammation: dual anti-inflammatory and pro-resolution lipid mediators. Nat Rev Immunol. 2008 May;8(5):349-61. doi: 10.1038/nri2294. PMID 18437155
- [Background] Colas RA, Shinohara M, Dalli J, Chiang N, Serhan CN. Identification and signature profiles for pro-resolving and inflammatory lipid mediators in human tissue. Am J Physiol Cell Physiol. 2014 Jul 1;307(1):C39-54. doi: 10.1152/ajpcell.00024.2014. Epub 2014 Apr 2. PMID 24696140
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Derived] Callan N, Hanes D, Bradley R. Early evidence of efficacy for orally administered SPM-enriched marine lipid fraction on quality of life and pain in a sample of adults with chronic pain. J Transl Med. 2020 Oct 21;18(1):401. doi: 10.1186/s12967-020-02569-5. PMID 33087142